CLINICAL TRIAL: NCT01379118
Title: Comparison of Clinical Scales and Quantitative Knee Motion Data in Assessing the Clinical Outcomes and Performance of Total Knee Replacement Patients Before and After Surgery
Brief Title: Comparison of Clinical Outcomes and Performance of Total Knee Replacement Patients Before and After Surgery
Acronym: TKR
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gary Botimer, M.D. and Chairman, Loma Linda University
Other Study IDs: 5110158
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Degenerative Joint Disease; Osteoarthritis; Knee Injury, Trauma; Connective Tissue Disorder; Pain; Loss of Function
Keywords: Total knee replacement
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Knee Injuries; Wounds and Injuries; Connective Tissue Diseases; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to determine the relevancy of clinical scales for outcome measures as compared to flexion angle and other gait measures. Clinical outcomes measures in the form of the Knee Society Score and the WOMAC Score will be obtained from patients. Gait data will also be obtained from total knee replacement (TKR) patients at pre-operative and post-operative times. Gait data will be measured on unaffected normal controls as a second baseline.

The hypothesis is that the subjects clinical outcome measures do not accurately reflect gait dependent outcomes amd functional performance of the total knee replacement.

DETAILED DESCRIPTION:
Patients scheduled to undergo unilateral total knee replacement (TKR) surgery will be the subjects of the study. A control group of Healthy volunteers, will serve as a control group. The control group will be matched as close as possible by age and gender to the TKR group. Both pre and post-operative (3 weeks, 6, 9 and 12 months follow-up) measurements will be performed on the TKR group.

A Intelligent Device for Energy Expenditure and Activity (IDEEA) will be used to record body motion, the sensors for the IDEEA device will be placed on the patient and secured with adhesive tape(if not allergic) once the IDEEA device is properly placed on the patient, measuring and calibrating can start.

The patient will be required to perform tasks, walking at a normal pace for approximately 100 feet on a level surface, walk up and down moderate incline ramp, climb stairs 7 to 8 steps, sit and rise from two chairs. Parameters will be measured on each subject, knee flexion angle( walking, stair climbing and sitting), velocity ( walking and stair climbing), Stride length (walking), Energy (walking, stair climbing, and sitting), other parameters will be added as needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* needs unilateral total knee replacement

Exclusion Criteria:

* Active infection
* Autoimmune disease/ parkinson's disease
* HIV
* psychosocial disorders that would preclude accurate evaluation or substance abuse
* allergic to
* pregnant
* active malignancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients that are healthy and patients that need a unilateral total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparison of Clinical Outcomes and Performance of Total Knee Replacement Patient before and after surgery | 36 months
  To determine the relevancy of clinical scales for outcome measures as compared to flexion angle and other gait measures. Clinical measures in the form of the Knee Society Score and the WOMAC Score will be obtained from patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gary D. Botimer, M.D., Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Healthcare, Deptartment of Orthopaedic Surgery, San Bernardino, California, United States